CLINICAL TRIAL: NCT06543719
Title: Safe Maximum Work Times and the Effectiveness of Work-rest Allocations in Mitigating Increases in Core Temperature During and on the Day Following Prolonged Heavy-Intensity Work in the Heat in Young and Older Workers
Brief Title: Initial Stay Times and Heat Mitigation Controls for Uncompensable Occupational Heat Stress - Part II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Principal investigator, University of Ottawa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2024-07
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Core Temperature; Heat Stress, Exertional; Heat Fatigue; Exercise
Keywords: Heat exposure; Heat strain; Body temperature; Thermoregulation; Occupational heat stress; Uncompensable heat stress; Aging
MeSH Terms: conditions — Heat Stress Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Younger adults. (Experimental): Adults aged 18-30 years with no pre-existing health conditions
  Interventions: Other: Simulated work in the heat
- Older adults. Adults aged 50-69 with no pre-existing health conditions (Experimental): Adults aged 50-69 with no pre-existing health conditions
  Interventions: Other: Simulated work in the heat

INTERVENTIONS:
Other: Simulated work in the heat — Participants perform a continuous heavy-intensity work bout (metabolic rate of ~260 W/m2) until core temperature reaches 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels), which is immediately followed by intermittent work using a 1:1 work-rest allocation, starting with a 30 min rest break followed by a 30 min work bout for a total work duration of ~240 min. The work protocol is performed in the morning of day 1, and repeated in a post-lunch work period (i.e., afternoon of day 1) and on the morning of the next day (i.e., morning of day 2).

SUMMARY:
Workplaces rely on upper heat stress limits provided by the American Conference of Governmental Industrial Hygienists (ACGIH) to manage the health and safety of workers in hot environments. This is primarily achieved by interspersing work with rest periods, the length of which is dictated by environmental conditions and work intensity, to maintain core temperature at or below 38.0°C (equivalent to a 1°C increase in body core temperature above resting levels). However, these guidelines employ a "one size fits all" approach to exposure limits that does not consider individual variation (e.g., age) between workers. Moreover, they fail to provide direction on the safe, initial stay times before these heat-mitigation controls should be employed (i.e., rest breaks) in conditions exceeding upper heat stress limits. While recent work has generated estimates of the initial stay times for young to older men before heat-mitigation controls are required for moderate-intensity work, information on initial stay times for heavy-intensity work remains to be assessed. This project will assess the initial stay times for heavy-intensity work for a single work bout as well as for a second work bout that is preceded by an extended rest period such as a lunch break and a work bout performed on the next day to determine if refinements in initial stay times across these periods may be required. Further, the investigators will evaluate if the application of recommended work-rest allocations thereafter would alleviate increases in core temperature for the duration of the work period (e.g., start of shift versus post-lunch period). Given the known age-differences in heat loss that can modulate core temperature regulation during an exercise-heat stress, the investigators will assess responses response in young and older adults.

ELIGIBILITY:
Inclusion Criteria:

* young (18-30 years) and older adults (50-69 years)
* habitually active, not endurance trained (<2 sessions per week, <150 minutes per week)
* non-smoking
* English or French speaking
* ability to provide informed consent

Exclusion Criteria:

* pre-existing health conditions (e.g., diabetes, hypertension)
* use of medication deemed to significantly modulate thermoregulatory function and heat tolerance (e.g., antidepressants, antihistamines, diuretics)
* engaged in jobs and/or activities that involve frequent exposure to hot environments (e.g., regular sauna use)

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Initial stay time | End of first (morning day 1) continuous work bout
  Total continuous work time to achieve an initial absolute increase in core temperature of 38°C (equivalent to a 1°C increase in body core temperature above resting levels) (note: in instances where a participant voluntarily terminates work prematurely before the absolute core temperature of ≥38°C (or relative increase of ≥1°C) is achieved or the absolute core temperature is <38°C (or relative increase of <1°C), the time of termination or end of the work bout will be taken as the initial stay time respectively).
Initial stay time | End of second (afternoon day 1) continuous work bout
  Total continuous work time to achieve an initial absolute increase in core temperature of 38°C (equivalent to a 1°C increase in body core temperature above resting levels) (note: in instances where a participant voluntarily terminates work prematurely before the absolute core temperature of ≥38°C (or relative increase of ≥1°C) is achieved or the absolute core temperature is <38°C (or relative increase of <1°C), the time of termination or end of the work bout will be taken as the initial stay time respectively).
Initial stay time | End of third (morning day 2) continuous work bout
  Total continuous work time to achieve an initial absolute increase in core temperature of 38°C (equivalent to a 1°C increase in body core temperature above resting levels) (note: in instances where a participant voluntarily terminates work prematurely before the absolute core temperature of ≥38°C (or relative increase of ≥1°C) is achieved or the absolute core temperature is <38°C (or relative increase of <1°C), the time of termination or end of the work bout will be taken as the initial stay time respectively).
Average core temperature | Period of work-rest allocations following initial stay time for morning day 1
  Average core temperature following initial stay time
Average core temperature | Period of work-rest allocations following initial stay time for afternoon day 1
  Average core temperature following initial stay time
Average core temperature | Period of work-rest allocations following initial stay time for morning of day 2
  Average core temperature following initial stay time

SECONDARY OUTCOMES:
Heart rate at initial stay time | End of first (morning day 1) continuous work bout
  Heart rate at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Heart rate at initial stay time | End of first (afternoon day 1) continuous work bout
  Heart rate at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Heart rate at initial stay time | End of first (morning day 2) continuous work bout
  Heart rate at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Average heart rate | Period of work-rest allocations following initial stay time for morning of day 1
  Average heart rate following initial stay time
Average heart rate | Period of work-rest allocations following initial stay time for afternoon of day 1
  Average heart rate following initial stay time
Average heart rate | Period of work-rest allocations following initial stay time for morning of day 2
  Average heart rate following initial stay time
Skin temperature at initial stay time | End of first (morning day 1) continuous work bout
  Skin temperature (4 sites) measured at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Skin temperature at initial stay time | End of first (afternoon day 1) continuous work bout
  Skin temperature (4 sites) measured at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Skin temperature at initial stay time | End of first (morning day 2) continuous work bout
  Skin temperature (4 sites) measured at the initial increase in absolute core temperature of 38°C (or relative increase of 1°C)
Average skin temperature | Period of work-rest allocations following initial stay time for morning of day 1
  Average heart rate following initial stay time
Average skin temperature | Period of work-rest allocations following initial stay time for afternoon of day 1
  Average heart rate following initial stay time
Average skin temperature | Period of work-rest allocations following initial stay time for morning of day 2
  Average heart rate following initial stay time
Systolic blood pressure | End of first (morning day 1) work period
  Arterial blood pressure measured via automated oscillometry
Systolic blood pressure | End of second (afternoon day 1) work period
  Arterial blood pressure measured via automated oscillometry
Systolic blood pressure | End of third (morning day 2) work period
  Arterial blood pressure measured via automated oscillometry
Diastolic blood pressure | End of first (morning day 1) work period
  Arterial blood pressure measured via automated oscillometry
Diastolic blood pressure | End of second (afternoon day 1) work period
  Arterial blood pressure measured via automated oscillometry
Diastolic blood pressure | End of third (morning day 1) work period
  Arterial blood pressure measured via automated oscillometry
Mean arterial pressure | End of first (morning day 1) work period
  Calculated as 1/3 * systolic blood pressure + 2/3 * diastolic blood pressure
Mean arterial pressure | End of second (afternoon day 1) work period
  Calculated as 1/3 * systolic blood pressure + 2/3 * diastolic blood pressure
Mean arterial pressure | End of third (morning day 2) work period
  Calculated as 1/3 * systolic blood pressure + 2/3 * diastolic blood pressure
Rate pressure product | End of first (morning day 1) work period
  Calculated as systolic blood pressure * heart rate
Rate pressure product | End of second (afternoon day 1) work period
  Calculated as systolic blood pressure * heart rate
Rate pressure product | End of third (morning day 2) work period
  Calculated as systolic blood pressure * heart rate
Fluid consumption | End of first (morning day 1) work period
  Cumulative fluid consumption calculated by weighing the participant's water intake
Fluid consumption | End of second (afternoon day 1) work period
  Cumulative fluid consumption calculated by weighing the participant's water intake
Fluid consumption | End of third (morning day 2) work period
  Cumulative fluid consumption calculated by weighing the participant's water intake
Fluid loss | End of first (morning day 1) work period
  Fluid loss calculated as the change in body mass (corrected for food/fluid consumption).
Fluid loss | End of second (afternoon day 1) work period
  Fluid loss calculated as the change in body mass (corrected for food/fluid consumption).
Fluid loss | End of third (morning day 2) work period
  Fluid loss calculated as the change in body mass (corrected for food/fluid consumption).
Change in plasma volume | End of first (morning day 1) work period
  Determined from venous blood samples
Change in plasma volume | End of second (afternoon day 1) work period
  Determined from venous blood samples
Change in plasma volume | End of third (morning day 2) work period
  Determined from venous blood samples
Thermal comfort scale | End of first (morning day 1) continuous work bout
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thermal comfort scale | End of second (afternoon day 1) continuous work bout
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thermal comfort scale | End of third (morning day 2) continuous work bout
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thermal comfort scale | Period of work-rest allocations following initial stay time for morning of day 1
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thermal comfort scale | Period of work-rest allocations following initial stay time for afternoon of day 1
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thermal comfort scale | Period of work-rest allocations following initial stay time for morning of day 2
  Thermal comfort assessed via a visual analog scale ("How comfortable does your body temperature feel?") (4: very uncomfortable to 1: comfortable)
Thirst sensation scale | End of first (morning day 1) continuous work bout
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Thirst sensation scale | End of second (afternoon day 1) continuous work period
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Thirst sensation scale | End of third (morning day 2) continuous work period
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Thirst sensation scale | Period of work-rest allocations following initial stay time for morning of day 1
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Thirst sensation scale | Period of work-rest allocations following initial stay time for afternoon day 2
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Thirst sensation scale | Period of work-rest allocations following initial stay time for morning of day 2
  Assessed via a visual analog scale ("How thirsty are you?") (9: very, very thirsty to 1: Not thirsty at all)
Rating of Perceived Exertion | End of first (morning day 1) continuous work bout
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Rating of Perceived Exertion | End of second (afternoon day 1) continuous work bout
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Rating of Perceived Exertion | End of third (morning day 2) continuous work bout
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Rating of Perceived Exertion | Period of work-rest allocations following initial stay time for morning of day 1
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Rating of Perceived Exertion | Period of work-rest allocations following initial stay time for afternoon of day 1
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Rating of Perceived Exertion | Period of work-rest allocations following initial stay time for morning of day 2
  Perceived exertion assessed via a self-report questionnaire upon verbal prompting (6: no exertion at all to 20: maximal exertion).
Orthostatic Intolerance Symptoms Assessment | End of first (morning day 1) continuous work bout
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort"
Orthostatic Intolerance Symptoms Assessment | End of second (afternoon day 1) continuous work bout
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort"
Orthostatic Intolerance Symptoms Assessment | End of third (afternoon day 1) continuous work bout
  Cumulative sum of scores on 6 questions asking participant to rank symptoms associated with orthostatic intolerance. All symptoms scored on a scale from 0 (none) to 10 (worst possible) and include feelings of: (1) "dizziness, lightheadedness, feeling faint, or feeling like you might black out"; (2) "Problems with vision (blurring, seeing spots, tunnel vision, etc.)"; (3) "Weakness"; (4) "Fatigue"; (5) "Trouble concentrating"; and (6) "Head and neck discomfort"

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada